CLINICAL TRIAL: NCT03940794
Title: Pelvic Floor Muscle Contraction in Response to Different Verbal Instructions in Women With Urinary Incontinence - A Self-controlled Clinical Trial
Brief Title: Pelvic Floor Muscle Contraction in Response to Different Verbal Instructions in Women With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ArielU
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence; Pelvic floor muscle contraction; Transabdominal ultrasound; Verbal instructions
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Single Group Assignment all participants will receive the same verbal instruction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verbal instruction (Experimental): The participants will be instructed to contract the pelvic floor muscle with the following verbal instruction: (1) "contract your pelvic floor - all sphincters"; (2) "contract your anus"; (3) "contract your pelvic floor as if you're trying to stop urinating".Those who will not be able to contract will be taught by the ultrasound as biofeedback.
  Interventions: Other: Verbal instruction

INTERVENTIONS:
Other: Verbal instruction — Verbal instruction for pelvic floor contraction will be given to participants. A transabdominal Ultrasound examination will be conducted to asses urinary bladder displacement being a marker for pelvic floor muscle function.
  Other Names: Trans abdominal Ultrasound examination for pelvic floor contraction

SUMMARY:
The aim of this study is to investigate which verbal instruction will lead to the most efficient contraction of pelvic floor muscles (PFM) in patients with urinary incontinence.

and to examine whether correct PFM contraction can be taught by transabdominal ultrasound, which is used as biofeedback.

Pelvic floor muscle contraction will be evaluated via transabdominal ultrasound.

DETAILED DESCRIPTION:
A self-controlled clinical trial is planned for patients who receive physiotherapy for pelvic floor rehabilitation at one of the Meuhedet Institutes' physiotherapy clinics.

Each participant will be asked to contract the pelvic floor muscles using three different verbal instructions: (1) "contract your pelvic floor - all sphincters"; (2) "contract your anus"; (3) "contract your pelvic floor as if you're trying to stop urinating". Those who will not be able to contract will be taught by the ultrasound as biofeedback.

The assessment of pelvic floor contraction will be measured by measuring bladder displacement via abdominal ultrasound. A curved linear array transducer will be placed in the transverse plane immediately suprapubically over the lower abdomen angled at 15-30 degrees from the vertical. An on-screen caliper and measurement tool will be used to measure bladder displacement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of urinary incontinence
* Understand the language and simple instruction
* Willing to participate in the study

Exclusion Criteria:

* Has been treated before for pelvic floor rehabilitation by a physiotherapist
* Received medication or surgery for the problem

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
urinary bladder displacement in millimeters during verbal instructions | baseline
  bladder displacement will be measured via diagnostic ultrasound using the on screen caliper tool

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | Baseline
  Questionnaire regarding symptoms of urinary incontinence,scale range 0-21 points.
  higher values represent worse outcome
Pelvic floor muscles endurance of contraction in seconds | Baseline
  time of muscle contraction will be measured during the last contraction in each instruction

CONTACTS AND LOCATIONS:
Overall Officials: Noa Ben Ami, PhD, Principal Investigator — Ariel University
Locations (1):
- Noa Ben Ami, Ariel, Israel

IPD SHARING:
Plan to Share IPD: No
the result of the study will be analyzed. a paper will be submitted to an international journal with study description including methods, examination protocol results.

REFERENCES:
- [Result] Ben Ami N, Dar G. What is the most effective verbal instruction for correctly contracting the pelvic floor muscles? Neurourol Urodyn. 2018 Nov;37(8):2904-2910. doi: 10.1002/nau.23810. Epub 2018 Aug 28. PMID 30152550
- [Result] Bo K, Sherburn M. Evaluation of female pelvic-floor muscle function and strength. Phys Ther. 2005 Mar;85(3):269-82. PMID 15733051
- [Result] Oliveira M, Ferreira M, Azevedo MJ, Firmino-Machado J, Santos PC. Pelvic floor muscle training protocol for stress urinary incontinence in women: A systematic review. Rev Assoc Med Bras (1992). 2017 Jul;63(7):642-650. doi: 10.1590/1806-9282.63.07.642. PMID 28977091